CLINICAL TRIAL: NCT04587037
Title: A Clinical Study Comparing Superior Capsule Reconstruction Using Fascia Lata Allograft With Human Dermal Allograft for Irreparable Rotator Cuff Tear
Brief Title: A Clinical Study Comparing Superior Capsule Reconstruction Using Different Graft for Irreparable Rotator Cuff Tear
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Chunyan Jiang, Director of Sports Medicine Service of Beijing Jishuitan hospital, Beijing Jishuitan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CJiang-SCR Compare
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Rotator Cuff Tears
Keywords: Irreparable Rotator Cuff Tears; Superior Capsular Reconstruction; Fascia lata allograft; human dermal allograft
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascia lata group (Experimental)
  Interventions: Procedure: fascia lata allograft
- Dermal allograft group (Experimental)
  Interventions: Procedure: human dermal allograft

INTERVENTIONS:
Procedure: fascia lata allograft — underwent superior capsule reconstruction using fascia lata allograft
  Arms: Fascia lata group
Procedure: human dermal allograft — underwent superior capsule reconstruction using human dermal allograft
  Arms: Dermal allograft group

SUMMARY:
Biomechanical and clinical success of the superior capsule reconstruction (SCR) using fascia lata (FL) grafts has been reported in treating irreparable rotator cuff tear. Human dermal (HD) allograft has been used successfully for SCRs; however, the clinical comparative study between FL and HD have not been reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients with irreparable rotator cuff tears
* Underwent superior capsule reconstruction using fascia lata allograft with human dermal allograft
* At least two years follow-up

Exclusion Criteria:

* reparable rotator cuff tears
* underwent partial repair or reverse total shoulder arthroplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) score | 2 year postoperatively
  A patient-reported outcome measurement
Acromiohumeral distance (AHD) | 1 year postoperatively
  measured in X-ray
Retear rate | 1 year postoperatively
  Measured in MRI

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Jiang, Principal Investigator — Sports Medicine Service, Beijing Jishuitan hospital

IPD SHARING:
Plan to Share IPD: No